CLINICAL TRIAL: NCT06736678
Title: Efficacy of Oral Immunonutrition Therapy in Reducing Acute Toxicity After Neoadjuvant Chemoradiotherapy Among Pancreatic Cancer Patients: a Prospective, Single-arm Clinical Trial
Brief Title: Oral Immunonutrition Therapy to Reduce Acute Toxicity After Neoadjuvant Chemoradiotherapy Pancreatic Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, WeiWei Xiao, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B2023-360-01
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Cancer; Neoadjuvant Chemoradiotherapy; Immunonutrition
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Immunonutrition Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Dietary Supplement: Oral Immunonutrition

INTERVENTIONS:
Dietary Supplement: Oral Immunonutrition — Patients receive enteral immunonutrition, Oral Impact® Nestle for 6 weeks from one week before radiotherapy;

SUMMARY:
A prospective, single-arm clinical trial is conducted to investigate the role of oral immunonutrion in reducing acute toxicity after neoadjuvant chemoradiotherapy among pancreatic cancer patients.

DETAILED DESCRIPTION:
Pancreatic cancer has a poor prognosis for its high malignancy. Radical surgical resection is an effective means for prolonging survival. However, only a few patients can be directly treated with surgical resection. Neoadjuvant therapy can reduce the tumor size, improve the relationship between the tumor and adjacent blood vessels，to gain surgical opportunities and prolonging patients' survival.

Nutritional treatment of cancer has been valued by more and more researchers. As an important branch of nutrition therapy, immunonutrition plays an important role in regulating the immune. Studies have shown that immunonutrition can reduce antitumor treatment related toxicity among patients with head and neck cancer, esophageal cancer. At present, most studies on immunonutrition therapy focus on perioperative patients, and there is no study on patients with pancreatic cancer undergoing radiotherapy.

This prospective, single-arm clinical trial aimed to explore the efficacy and safety of oral immunonutrition therapy in reducing acute toxicity after neoadjuvant chemoradiotherapy among pancreatic cancer patients. A total of 98 pancreatic cancer patients will be enrolled. All of the patients will receive oral immunonutrition therapy for 6 weeks from one week before radiotherapy. The total follow time is 4 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathologically confirmed pancreatic ductal epithelial malignant tumors;
* 2. Resectable pancreatic cancer treated with neoadjuvant chemoradiotherapy, or nonresectable locally advanced pancreatic cancer treated with neoadjuvant or radical chemoradiotherapy;
* 3.Nutritional Risk Screening 2002 (NRS2002) ≥3 and Patient-Generated Subjective Global Assessment (PG-SGA) performance status B;
* 4. Age 18 years and older;
* 5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* 6. Expected survival time more than 3 months;
* 7. History of antineoplastic therapy;

Exclusion Criteria:

* 1. Known allergy or intolerance to any component of investigational Oral Immunonutrition;
* 2. History of Oral Immunonutrition use within one month prior to enrollment;
* 3. Tumor compresses the major duodenal papilla, and /or appeared jaundice, acute pancreatitis;
* 4. Patients with contraindications for antineoplastic therapy, such as coronary heart disease, cerebral infarction, cerebral hemorrhage or other serious diseases;
* 5. Liver, kidney and blood coagulation function failure;
* 6. Patients with hemopathy;
* 7. Patients with active infections;
* 8. Patients with other primary tumor;
* 9. Patients with other medical diseases that seriously affected nutritional status;
* 10.Subjects deemed by the investigator have other factors that may be ineligible for enrollment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of grade 3 or higher acute toxicity related to neoadjuvant chemoradiotherapy | Baseline, week 17
  Grading of acute toxicity would be assessed according to National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

SECONDARY OUTCOMES:
Usual Body Weight Percentage(UBW%) | Baseline, Week 3,5,7,9,13,17
  The baseline weight would be considered as usual body weight. UBW%= current weight/usual weight ×100%
Nutritional Assessment | Baseline, Week 3,5,7,9,13,17
  Patient-Generated Subjective Global Assessment（PG-SGA）
Nutritional Risk | Baseline, Week 3,5,7,9,13,17
  Nutritional Risk Screening 2002 (NRS 2002)
Quality of Life | Baseline, Week 3,5,7,9,13,17
  The European Organisation for Research and Treatment of Cancer quality of life (EORTC QLQ-C30)
Inflammatory Indexes | Baseline; Week 7;
  The serum level of procalcitonin (PCT),C-reactive protein(CRP) , serum amyloid A(SAA).
Immunological Indexes | Baseline; Week 7;
  The white blood cell (WBC) count and neutrophil (NE) count.
Disease Control Rate (DCR) | Baseline; Week 13,17;
  Disease control rate (DCR) was defined as the percentage of CR+PR+SD among the patients who could be evaluated for efficacy.
Resectable Status Rate | Baseline; Week 13,17;
  Incidence rate of conversion from unresectable to resectable status after radiotherapy.
  Resectable status was defined according to the National Comprehensive Cancer Network (NCCN) Guidelines Version 1 2012. Tumors considered resectable were defined by the following objective criteria: (1) no distant metastases, (2)venous involvement of the portal vein demonstrating tumor abutment with impingement and narrowing of the lumen, encasement of the superior mesenteric vein (SMV)/portal vein allowing for safe resection and reconstruction, (3) no extension to the celiac axis, (4) tumor abutment of the SMA not to exceed >180° of the circumference of the vessel wall.
Radiotherapy Interruption (RTI) | Week 3,5,7,9;
  Radiotherapy interruption (RTI) often occurs because of severe acute treatment-related toxicity, disease progression, and patients' treatment compliance. RTI was defined as the difference between radiation treatment time and planned radiation time.
Overall Survival (OS) | Week 17; Year 2;
  Overall survival was calculated from the date of treatment to either the date of death or last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Xiao, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China